CLINICAL TRIAL: NCT05407961
Title: A Phase 1b, 2-Part, Investigator- and Participant-Blind, Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY3532226 in Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3532226 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17835; 2021-003257-31 (EudraCT Number); J2V-MC-GZLB (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- LY3532226 + Dulaglutide (Part A) (Experimental): LY3532226 administered subcutaneously (SC) followed by dulaglutide administered SC.
  Interventions: Drug: LY3532226; Drug: Dulaglutide
- Placebo + Dulaglutide (Part A) (Placebo Comparator): Placebo administered SC followed by dulaglutide administered SC.
  Interventions: Drug: Placebo; Drug: Dulaglutide
- Dulaglutide + Placebo (Part B) (Active Comparator): Dulaglutide administered SC in combination with placebo given SC.
  Interventions: Drug: Placebo; Drug: Dulaglutide
- LY3532226 + Dulaglutide (Part B) (Experimental): LY3532226 administered SC in combination with Dulaglutide given SC.
  Interventions: Drug: LY3532226; Drug: Dulaglutide
- LY3532226 + Placebo (Part B) (Experimental): LY3532226 administered SC in combination with placebo given SC.
  Interventions: Drug: LY3532226; Drug: Placebo

INTERVENTIONS:
Drug: LY3532226 — Administered SC.
  Arms: LY3532226 + Dulaglutide (Part A); LY3532226 + Dulaglutide (Part B); LY3532226 + Placebo (Part B)
Drug: Placebo — Administered SC.
  Arms: Dulaglutide + Placebo (Part B); LY3532226 + Placebo (Part B); Placebo + Dulaglutide (Part A)
Drug: Dulaglutide — Administered SC.
  Other Names: Trulicity
  Arms: Dulaglutide + Placebo (Part B); LY3532226 + Dulaglutide (Part A); LY3532226 + Dulaglutide (Part B); Placebo + Dulaglutide (Part A)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY3532226 in participants with type 2 diabetes mellitus (T2DM). Blood tests will be performed to check how much LY3532226 gets into the bloodstream and how long it takes the body to eliminate it. This is a 2-part study and will last approximately 16 weeks excluding screening period for each part, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes mellitus (T2DM) for at least 3 months before screening
* Have the following glycosylated hemoglobin (HbA1c) levels at screening:

  1. HbA1c >/= 7.0% to </= 10.0% for participants treated with diet and exercise alone and participants treated with metformin alone, and
  2. HbA1c >/= 6.0% to </= 9.5% for participants treated with dipeptidyl peptidase inhibitor-4 (DPP-4) (with/without metformin) inhibitors and participants treated with metformin and sodium-glucose cotransporter-2 (SGLT-2) inhibitor
* Participants treated with diet and exercise alone or on a stable dose of metformin for at least 3 months
* Participants with body weight up to 150 kilograms (kg) and body mass index (BMI) of 23.0 to 45.0 kilograms per meter squared (kg/m²)
* Male participants who agree to use effective methods of contraception and female participants not of childbearing potential

Exclusion Criteria:

* Participants who have uncontrolled diabetes defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to screening
* Have a clinically significant abnormality ECG
* Have obesity induced by other endocrine disorders such as Cushing's syndrome or Prader-Willi syndrome
* Are on any glucose-lowering medications other than metformin, SGLT-2 inhibitors and/or DPP4
* Have received chronic systemic glucocorticoid therapy (>2 weeks) in the past 6 months
* Have an average weekly alcohol intake that exceeds 21 units per week (males 65 years of age or lesser) and 14 units per week (females and males 65 years of age or older)
* Smoke more than 10 cigarettes, or cigarette equivalent, per day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 16
  A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module
Part B: Change from Baseline in Total Clamp Disposition Index (cDI) | Baseline up to Week 12
  Change from Baseline in Total cDI

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3532226 | Predose on Day 1 through Week 16
  PK: Cmax of LY3532226
Part A: PK: Area Under the Concentration Versus Time Curve (AUC) of LY3532226 | Predose on Day 1 through Week 16
  PK: AUC of LY3532226
Part B: Change from Baseline in Insulin Secretion Rate (ISR) from hyperglycaemic clamp | Baseline through Week 12
  Change from Baseline in ISR from hyperglycaemic clamp
Part B: Change from Baseline in β-cell Glucose Sensitivity (GS) from hyperglycaemic clamp | Baseline through Week 12
  Change from Baseline in β-cell GS from hyperglycaemic clamp
Part B: Change from Baseline in Hyperinsulinemic Euglycemic Clamp M-value | Baseline through Week 12
  Change from Baseline in Hyperinsulinemic Euglycemic Clamp M-value
Part A & B: Change from Baseline in Fasting and Post meal Glucose during Standardized Mixed-meal Tolerance Test (sMMTT) | Baseline through Week 16
  Change from Baseline in Fasting and Post meal Glucose during sMMTT
Part A & B: Change from Baseline in Glycosylated Haemoglobin (HbA1c) | Baseline through Week 16
  Change from Baseline in HbA1c
Part A & B: Change from Baseline in Glucagon Concentration at Fasting and Post meal during sMMTT | Baseline through Week 16
  Change from Baseline in Glucagon Concentration at Fasting and Post meal during sMMTT

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No